CLINICAL TRIAL: NCT02745782
Title: A Study of the Trigeminal Cardio-Reflex in Endodontic and Other Dental Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: YI SHENG HUANG (Other)
Responsible Party: Sponsor-Investigator, YI SHENG HUANG, Professor, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Other Study IDs: CS 14112
Record Dates: First submitted 2016-04-09; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Pulpitis
Keywords: Pulpitis; Syncope; Trigeminal Cardio-Reflex
MeSH Terms: conditions — Pulpitis; Syncope | interventions — Observation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational Study — Observational Study

SUMMARY:
This study sought to comprehend the relationship between syncope and dental related therapy. If the relationship between dental related therapies and syncope is proved, clinical dentists will be remained to monitor changes of patient's blood pressure during root canal procedure.

DETAILED DESCRIPTION:
This study sought to comprehend the relationship between syncope and dental related therapy. If the relationship between dental related therapies and syncope is proved, clinical dentists will be remained to monitor changes of patient's blood pressure during root canal procedure.

Previous Trigemino-Cardiac Reflex(TCR) related studies reported that stimulation of trigeminal nerve induces trigeminal nerve reflection, and then causes blood pressure rapidly decreasing. Finally, sudden blood pressure decreasing results in syncope. Clinical data has been collected and analyzed in the past four months, and the primary results showed significantly difference. This phenomenon may be probably observed in other dental treatments. Hence, the objective of this study is to remind clinical dentists to monitor patients' physical conditions when conducting root canal relevant treatments and to avoid situations such as syncope, and reduce medical disputes and benefit dentists and patient as a result. In the recent year, syncope often occurs during denture procedures. The value of this study will inform clinical dentist to notice risk of dental relative treatments. In addition, it will improve patients' safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the informed consent forms
* Patients with Pulpitis
* Patients aged 20 or order

Exclusion Criteria:

* Patients aged under 20

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators collected data from adult patients who agreed to participate in the study and accepted relevant treatments including filling, extraction, scaling, implant, and crown bridge preparation (no more than 500 patients in each treatment item) before September 2016. Previous studies shows that TCR is more often happen in young patients. Therefore, to avoid ethical issue, adult patients are more suitable in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Blood Pressure(MABP) lower than 20% | Through routine dental treatment completion, an average of 1 hour
Heart Rate (HR): lower than 60 beats/ minute | Through routine dental treatment completion, an average of 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Tsui Hsien Huang, Ph.D, Principal Investigator — CSMU
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schipke JD, Cleveland S, Caspers C. Computer-assisted paranasal sinus operation induces diving bradycardia. Am J Otolaryngol. 2013 Jul-Aug;34(4):353-4. doi: 10.1016/j.amjoto.2012.12.004. Epub 2013 Jan 14. PMID 23332411
- [Background] Yorgancilar E, Gun R, Yildirim M, Bakir S, Akkus Z, Topcu I. Determination of trigeminocardiac reflex during rhinoplasty. Int J Oral Maxillofac Surg. 2012 Mar;41(3):389-93. doi: 10.1016/j.ijom.2011.12.025. Epub 2012 Jan 11. PMID 22240287
- [Background] Bohluli B, Ashtiani AK, Khayampoor A, Sadr-Eshkevari P. Trigeminocardiac reflex: a MaxFax literature review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Aug;108(2):184-8. doi: 10.1016/j.tripleo.2009.03.050. PMID 19615657
- [Background] Lubbers HT, Zweifel D, Gratz KW, Kruse A. Classification of potential risk factors for trigeminocardiac reflex in craniomaxillofacial surgery. J Oral Maxillofac Surg. 2010 Jun;68(6):1317-21. doi: 10.1016/j.joms.2009.12.039. Epub 2010 Mar 29. PMID 20347202
- [Background] Schaller B, Probst R, Strebel S, Gratzl O. Trigeminocardiac reflex during surgery in the cerebellopontine angle. J Neurosurg. 1999 Feb;90(2):215-20. doi: 10.3171/jns.1999.90.2.0215. PMID 9950491